CLINICAL TRIAL: NCT03367806
Title: Caffeine Consumption and Mortality in Diabetes: an Analysis of National Health and Nutrition Examination Survey (NHANES) 1999-2010
Brief Title: Caffeine Consumption and Mortality in Diabetes
Status: Completed | Type: Observational
Sponsor: João Sérgio Neves (Other)
Responsible Party: Sponsor-Investigator, João Sérgio Neves, MD, Universidade do Porto
Organization: Universidade do Porto (Other)
Other Study IDs: Caffeine-DM
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous studies suggested an inverse relationship between coffee consumption and mortality in the general population. Furthermore, an inverse association between coffee consumption and serum biomarkers of inflammation and insulin resistance has been described. Prospective studies showed that coffee consumption might be associated with reduction in the incidence of type 2 diabetes. Although caffeine consumption appears to be associated with a decreased risk of developing type 2 diabetes, the relationship between caffeine consumption and mortality in patients with diabetes remains uncertain. The current analysis aimed to assess the effects of caffeine consumption and caffeine source on all-cause, cardiovascular and cancer mortality among patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* NHANES participants from 1999 to 2010 above 18-year old, with diagnosis of diabetes

Exclusion Criteria:

* Implausible alimentary reports (defined as consumption of less than 500 kcal/day or more than 3500 kcal/day)
* Missing information on caffeine consumption
* Missing information on mortality

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: NHANES is a nationally-representative, cross-sectional study of nutrition and health for individuals residing in the U.S.
Sampling Method: Probability Sample
Enrollment: 3052 (Actual)
Dates: Start 1999-01 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | From baseline until death or censoring on 31 December 2011, whichever came first, assessed up to 12 years
  All-cause mortality as assessed by NHANES linked National Death Index public-access

SECONDARY OUTCOMES:
Cardiovascular mortality | From baseline until death or censoring on 31 December 2011, whichever came first, assessed up to 12 years
  Cardiovascular mortality as assessed by NHANES linked National Death Index public-access
Cancer mortality | From baseline until death or censoring on 31 December 2011, whichever came first, assessed up to 12 years
  Cancer mortality as assessed by NHANES linked National Death Index public-access